CLINICAL TRIAL: NCT06880211
Title: Activity Snippets for Sustainable Promotion of Physical Activity in Everyday Working Life - a Randomized Controlled Trial
Brief Title: Activity Snippets for Sustainable Promotion of Physical Activity in Everyday Working Life (ActivitySnippets)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Niederrhein University of Applied Sciences (Other)
Collaborators: Deutsche Sporthochschule Köln (Other)
Responsible Party: Principal Investigator, Lukas Streese, Dr. sc. med., Niederrhein University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 054/2025
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Physical Inactivity
Keywords: Physical Inactivity; Bus driver; Tram driver; activity snippets; Promotion of physical activity; Company health management
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to an intervention group or a control group. The intervention group will receive activity snippets for 16 weeks. The control group will receive WHO recommendations for physical activity.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physical activity recommendations (Active Comparator): The control group will receive the latest World Health Organization recommendations for physical activity for 16 weeks.
  Interventions: Other: physical activity recommendations
- activitysnippets (Experimental): The intervention group will receive a set of activity snippets for 16 weeks, consisting of a series of short exercises designed to improve muscle strength, increase physical activity levels at work and reduce stress.
  Interventions: Other: activitysnippets

INTERVENTIONS:
Other: physical activity recommendations — The participants (bus and tram drivers) in the control group will receive the latest World Health Organization recommendations for physical activity in written form.
  Arms: physical activity recommendations
Other: activitysnippets — Participants (bus and tram drivers) in the intervention group will receive the ActivitySnippets toolbox. The toolbox was developed through collaborative workshops with the target group, sports scientists and physiotherapists to create a sustainable, occupation-specific and evidence-based physical activity promotion. The toolbox, which provides simple incentives to integrate physical activity into everyday working life, consists of 30 to 40 activity snippets (exercise cards). The design of the toolbox allows for individualization and variation of the exercise cards. The aim of the exercises is to improve muscle strength, increase physical activity levels at work and reduce stress. All exercises can be performed for between 10 and 60 seconds, allowing for realistic implementation in everyday working life. Participants are encouraged to incorporate the exercises into their daily work routine as often as possible.
  Arms: activitysnippets

SUMMARY:
The ActivitySnippets study will investigate the effects of short activity snippets on the sedentary behavior of bus and tram drivers. The main research question is: Do activity snippets increase the amount of time bus and tram drivers spend in a physically active state and reduce the amount of sedentary time during working hours? This research question will be investigated with a randomized controlled trial.

DETAILED DESCRIPTION:
Physical inactivity is a global health burden and a major risk factor for noncommunicable diseases, which imposes a significant economic burden on health systems (Polo-López et al., 2024). On average, adults spend between 50 and 60% of their waking hours in sedentary behavior, with prolonged sitting significantly associated with increased all-cause mortality (Varela-Mato et al., 2015). Bus and tram drivers are particularly affected, spending up to 12 hours per day sitting, while also being exposed to work-related risk factors such as poor posture and strict schedules (Brodie et al., 2021; Varela-Mato et al., 2015).

Despite the availability of numerous health-promoting interventions for office workers, there is a lack of specialized, evidence-based health-promoting interventions tailored to the specific needs of bus and tram drivers. Research suggests that even short and low intensity physical activity can have health benefits (Koemel et al., 2024).

This research project aims to address the existing research gap by evaluating the effectiveness of short, simple and practical 'activity snippets' in reducing occupational physical inactivity among bus and tram drivers through a randomized controlled trial. Specifically, the study will investigate whether the implementation of activity snippets leads to a significant redistribution of sedentary time towards more active behavior compared to current World Health Organization (WHO) recommendations for physical activity.

A total of 75 bus and tram drivers from "Stadtwerke Krefeld", a public transport company in North Rhine-Westphalia (Germany), will be recruited to participate. At baseline, participants will wear an activity tracker for 10 days to measure acceleration, heart rate and other relevant parameters. Standardized and validated methods will be used to assess body composition, physical activity levels, strength and mobility. Participants will then be randomly assigned to either the intervention or control group.

The intervention group will receive a set of activity snippets for 16 weeks, consisting of a series of short exercises designed to improve muscle strength, increase activity levels at work and reduce stress. The control group will receive the latest WHO recommendations for physical activity. Throughout the intervention period, the research team will provide regular telephone support to ensure adherence, and both groups will wear an activity tracker for 10 days. Following the 16-week intervention, all baseline measures will be repeated, and user experience and acceptability of the activity snippets will be assessed. At the end of the study, participants in the control group will also be given access to the activity snippets. To assess potential long-term effects, a voluntary follow-up assessment, including 10 days of activity tracking, will be conducted three months after the end of the study.

This study aims to provide robust scientific evidence on the effectiveness of activity snippets in reducing prolonged sedentary time and increasing physical activity, and to assess their feasibility in the everyday working lives of bus and tram drivers. In addition, the findings could provide a basis for wider implementation in other inactive occupational groups. Ultimately, this research contributes to the advancement of both occupational and public health promotion strategies and supports the development of sustainable, evidence-based workplace interventions.

ELIGIBILITY:
Inclusion criteria:

* men and women
* Employees who are actively working as bus or tram drivers for the company "Stadtwerke Krefeld".

Exclusion criteria:

* Persons who work in other areas of the company "Stadtwerke Krefeld".
* Persons who are not actively employed as bus and/or tram drivers.
* Bus and/or tram drivers employed by other companies or subcontractors
* Persons who have not agreed in writing to take part in the study.
* Persons who have not signed the loan agreement for the activity tracker.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-03-19 (Actual); Primary Completion 2026-02-07 (Actual); Study Completion 2026-02-07 (Actual)

PRIMARY OUTCOMES:
The additional effect of short activity snippets, integrated into the daily work routine of bus and tram drivers, on the physical activity behavior compared to general physical activity recommendations. | From enrollment to the end of the 16 weeks intervention phase.
  Physical activity behavior will be quantified with the MATRIX ACTIVITY MONITOR, an activity tracker from Parmay Tech. This tracker will investigate the physical activity behavior for 7 days at each time point.

SECONDARY OUTCOMES:
The additional effect of short activity snippets, integrated into the daily work routine of bus and tram drivers, on daily steps compared to general physical activity recommendations. | From enrollment to the end of the 16 weeks intervention phase.
  Daily steps will be measured with the MATRIX ACTIVITY MONITOR, an activity tracker from Parmay Tech. This tracker will investigate the physical activity behavior for 7 days at each time point.
The additional effect of short activity snippets, integrated into the daily work routine of bus and tram drivers, on muscular strength compared to general physical activity recommendations. | From enrollment to the end of the 16 weeks intervention phase.
  Muscular strength will be measured with an isometric force measurement device from SAUTER. The maximal Power of the upper (musculus biceps brachii) and lower (musculus quadriceps femoris) extremities will be measured.
The additional effect of short activity snippets, integrated into the daily work routine of bus and tram drivers, on flexibility compared to general physical activity recommendations. | From enrollment to the end of the 16 weeks intervention phase.
  A goniometer will be used to measure the flexibility of the spine and lower extremity during rotation and flexion.
The additional effect of short activity snippets, integrated into the daily work routine of bus and tram drivers, on perceived stress compared to general physical activity recommendations. | From enrollment to the end of the 16 weeks intervention phase.
  The perceived Stress Scale (PSS-10) will be used to quantify psychological stress.
The additional effect of short activity snippets, integrated into the daily work routine of bus and tram drivers, on helth-related quality of life compared to general physical activity recommendations. | From enrollment to the end of the 16 weeks intervention phase.
  The Short Form Health Survey (SF-12), a self-reported questionnaire, will be used to quantify health-related quality of life.
The additional effect of short activity snippets, integrated into the daily work routine of bus and tram drivers, on job satisfaction and work engagement compared to general physical activity recommendations. | From enrollment to the end of the 16 weeks intervention phase.
  The Copenhagen Psychosocial Questionnaire (COPSOQ) will be used to quantify self-reported job satisfaction and work engagement.
The additional effect of short activity snippets, integrated into the daily work routine of bus and tram drivers, on self-reported physical activity compared to general physical activity recommendations. | From enrollment to the end of the 16 weeks intervention phase.
  The Global Physical Activity Questionnaire will be used to quantify self-reported scale of physical activity. This questionnaire has 16 questions about intensity, frequency and duration in the domains of physical activity at work and leisure.
The additional effect of short activity snippets, integrated into the daily work routine of bus and tram drivers, on muscular and skeletal disorders compared to general physical activity recommendations. | From enrollment to the end of the 16 weeks intervention phase.
  An adapted questionnaire (MSB) will be used to analyze muscular and skeletal disorders; covering 9 body regions, 4-week prevalence, intensity and limitations in work or leisure.

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Streese-Schüler, Dr. sc. med., Principal Investigator — Niederrhein University of Applied Sciences
Locations (1):
- Hochschule Niederrhein, University of Applied Sciences, Krefeld, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request, selected study data will be shared.

REFERENCES:
- [Result] Polo-Lopez A, Calatayud J, Lopez-Bueno L, Nunez-Cortes R, Andersen LL, Lopez-Bueno R. Dose-response association of an accelerometer-measured physical activity with all-cause mortality and cardiovascular disease incidence: Prospective cohort with 76,074 participants. Prog Cardiovasc Dis. 2024 Nov-Dec;87:2-7. doi: 10.1016/j.pcad.2024.10.004. Epub 2024 Oct 9. PMID 39389333
- [Result] Brodie A, Pavey T, Newton C, Sendall MC. Australian bus drivers' modifiable and contextual risk factors for chronic disease: A workplace study. PLoS One. 2021 Jul 29;16(7):e0255225. doi: 10.1371/journal.pone.0255225. eCollection 2021. PMID 34324584
- [Result] Koemel NA, Ahmadi MN, Biswas RK, Koster A, Atkin AJ, Sabag A, Stamatakis E. Can incidental physical activity offset the deleterious associations of sedentary behaviour with major adverse cardiovascular events? Eur J Prev Cardiol. 2025 Jan 6;32(1):77-85. doi: 10.1093/eurjpc/zwae316. PMID 39325719
- [Result] Varela-Mato V, Yates T, Stensel DJ, Biddle SJ, Clemes SA. Time spent sitting during and outside working hours in bus drivers: A pilot study. Prev Med Rep. 2015 Dec 3;3:36-9. doi: 10.1016/j.pmedr.2015.11.011. eCollection 2016 Jun. PMID 26844184